CLINICAL TRIAL: NCT05133583
Title: Effect of Laughter Yoga Therapy on Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Lokman Hekim University, Adiyaman University Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: lokman hekim
Record Dates: First submitted 2021-11-13; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervatonal (Experimental)
  Interventions: Other: Laughter yoga
- control (No Intervention)

INTERVENTIONS:
Other: Laughter yoga — The experimental group was interviewed in an online meeting prepared by a certified LY trainer.
  She received LY exercises once a week (40 minutes per session) for 6 weeks (6 sessions). Each The meeting was organized with a maximum of 12 people.
  Arms: intervatonal

SUMMARY:
Laughter yoga sessions, stretches and stretches, songs, clapping and body It starts with light warm-up techniques that include movements. These are to break down all kinds of inhibitions and It is aimed at developing the feelings of childlike play. breathing exercises lungs they are ready to laugh and are combined with the following series of laughing exercises. LY In order to provide group dynamics in therapy, the group should consist of at least 5-12 people.

provided. Real laughter is often experienced during laughter meditation; it's contagious and may trigger laughter in other people in the group, hence the group can establish greater connections with its members. Laughter yoga sessions are always held at the same time and in the same place to encourage the participation of individuals.

has been done.

DETAILED DESCRIPTION:
Laughter yoga sessions, stretches and stretches, songs, clapping and body It starts with light warm-up techniques that include movements. These are to break down all kinds of inhibitions and It is aimed at developing the feelings of childlike play. breathing exercises lungs they are ready to laugh and are combined with the following series of laughing exercises. LY In order to provide group dynamics in therapy, the group should consist of at least 5-12 people.

provided. Real laughter is often experienced during laughter meditation; it's contagious and may trigger laughter in other people in the group, hence the group can establish greater connections with its members. Laughter yoga sessions are always held at the same time and in the same place to encourage the participation of individuals.

has been done. Therapy sessions are between 40-45 minutes. Sessions started on time and was completed on time. In the research, a total of 6 sessions of laughter, once a week, yoga was done. The experimental group was interviewed in an online meeting prepared by a certified LY trainer.

She received LY exercises once a week (40 minutes per session) for 6 weeks (6 sessions). Each The meeting was organized with a maximum of 12 people.

ELIGIBILITY:
Inclusion Criteria:

* have a healthy baby

Exclusion Criteria:

* Absence of a psychiatric illness No chronic disease The newborn has no health problems

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women who have baby
Enrollment: 104 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Effect of Laughter Yoga therapy on postpartum Depression | 6 week
  The experimental group was interviewed in an online meeting prepared by a certified LY trainer.
  She received LY exercises once a week for 6 weeks (6 sessions). Each The meeting was organized with a maximum of 12 people. LY exercises were done as follows; Before starting the exercise, clapping-warm-up exercises for 10 minutes, deep breathing exercises were applied. The remaining 30 minutes were devoted to childlike acting and laughing exercises.
  Participants mainly focused on mind control, breathing control and relaxation body movements.
  they focused. Focusing on the emerging moment is a way to release negative emotions.
  It is assumed to provide temporary relief from negative thoughts while providing opportunities for

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Simsek Kucukkelepce, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided